CLINICAL TRIAL: NCT06253234
Title: Phase I Clinical Trial of Personalized Dendritic Cell Injection ZSNeo-DC1.1 in the Treatment of Recurrent or Progressive High-grade Glioma
Brief Title: Safety and Efficacy Study for DC Vaccine in Recurrent or Progressive High-grade Gliomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: ZhongSheng BioTech Inc. (Unknown)
Responsible Party: Principal Investigator, Yang Zhang, Clinical Professor, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSKY2023-1002
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: WHO Grade III Gliomas; WHO Grade IV Gliomas
MeSH Terms: interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Intervention Model Description: To evaluate the safety and tolerance of personalized DC vaccine in in recurrent or progressive high-grade gliomas.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Sequence A (Experimental)
  Interventions: Biological: personalized dendritic cell injection ZSNeo-DC1.1
- Treatment Sequence B (Experimental)
  Interventions: Biological: personalized dendritic cell injection ZSNeo-DC1.1

INTERVENTIONS:
Biological: personalized dendritic cell injection ZSNeo-DC1.1 — Sequence A: For the first 3 cycles, 1 week as a dosing cycle, the next 3 cycles, 3 weeks as a dosing cycle, a total of 6 dosing cycles Sequence B: For the first 3 cycles, 1 week as a dosing cycle, the next 3 cycles, 2 weeks as a dosing cycle, a total of 6 dosing cycles
  Other Names: DC vaccine

SUMMARY:
This is a single-center, open-label, multi-dose phase I clinical trial evaluating the safety, tolerability, and preliminary efficacy of ZSNeo-DC1.1, a personalized dendritic cell injection, in subjects with recurrent or progressive WHO grade III-IV gliomas post-standard treatment. The subjects are adult GBM patients who have undergone surgical resection for recurrence. After the completion of reoperation, subjects will receive autologous DC vaccine treatments as scheduled. The autologous genetic-modification-free DC cells will be loaded with multiple tumor neoantigen peptides and administered (i.h) to subjects. After 3 injections, the investigator will review subject's tolerance and compliance. The DLT observation period spans from the initial injection to 21 days after the third injection, aligning with the activation of anti-tumor immune response.

About 15 subjects will be enrolled. The study utilizes a fixed dose of 1×10^7 cells per injection and employs two immunization schedules A or B.

The trial is conducted in two stages:

Dose Confirmation Stage:

Enrollment of six subjects with recurrent or progressive gliomas following standard treatment. Each subject receives six subcutaneous injections of ZSNeo-DC1.1. Utilization of a standard "3+3" design for fixed dose confirmation and exploration of immunization schedules A and B.

Dose Expansion Stage:

Enrollment of at least six subjects with recurrent or progressive gliomas post-standard treatment. Administration of six subcutaneous injections of ZSNeo-DC1.1 to each subject, further investigating the safety and preliminary efficacy of ZSNeo-DC1.1 injection.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all the following criteria to be eligible:

  1. Age from 18 to 75 years (including 18 and 75 years old).
  2. Subjects with histologically or cytologically confirmed WHO grade III-IV gliomas experiencing recurrence or progression after standard treatment.
  3. Bridging therapy is allowed during the preparatory period after sample collection, with discontinuation at least 7 days or 5 drug half-lives (whichever is longer) before the initial treatment.
  4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2.
  5. Laboratory test results defining satisfactory hematological and organ function:

     Platelets (PLT) ≥ 90 × 10^9/L; Absolute Neutrophil Count (ANC) ≥ 1.5 × 10^9/L; Haemoglobin (HGB) ≥ 90 g/L; Serum Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5× ULN; Total Bilirubin (TBIL) ≤ 2.5 × ULN; Albumin (ALB) ≥ 3 g/dl; Creatinine clearance rate (CrCl) ≥ 45 mL/minute or Serum Creatinine ≤ 1.5 ×ULN; International Normalized Ratio (INR), Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN; Lipase ≤ 1.5 × ULN; Amylase ≤ 1.5 × ULN; Alkaline Phosphatase (ALP) ≤ 2.5 × ULN.
  6. Adequate tumor and blood samples for NGS gene sequencing can be obtained through tumor reduction surgery or biopsy. Peripheral blood mononuclear cell function is normal.
  7. Relief of any acute, clinically significant treatment-related toxicities (excluding alopecia) to ≤ Grade 1 before the first treatment.
  8. Heart function: Stable hemodynamics, LVEF ≥ 50%.
  9. Adequate venous access for PBMC collection, with no contraindications.
  10. Non-surgically sterilized reproductive-age subjects must use contraception during the study and have a negative pregnancy test.
  11. Expected survival period > 3 months.
  12. Voluntary participation, signed informed consent.
  13. Based on health and lab assessments, the investigator sees favorable risk-benefit for the subject in the clinical trial.
  14. Subjects must consistently comply, actively participate in follow-up visits, and undergo regular testing and evaluation at the research center throughout the trial.

Exclusion Criteria:

* Subjects meeting any of the following criteria are ineligible:

  1. Recent participation in other drug trials, concurrent anti-tumor therapy (excluding allowed bridging therapy) within 4 weeks before initial treatment, had blood transfusions, EPO, G-CSF, or GM-CSF in the 14 days before peripheral blood mononuclear cell collection, or received live virus vaccinations within 28 days before the first treatment.
  2. Subjects who had camptothecin sustained-release agent implantation surgery within 6 months before the initial treatment.
  3. Active autoimmune diseases, prolonged use of immunosuppressive therapy, or known egg allergy.
  4. Positive for HIV or syphilis antibodies, or active hepatitis B or C.
  5. Recent systemic immunosuppressive treatment within 30 days before the initial treatment.

     Note: Short-term, systemic immunosuppressive treatment may be considered in consultation with the investigator and sponsor approval. The washout period and its duration before the initial treatment will be decided in consultation with the sponsor for these patients.

     Allowed: Inhaled glucocorticoids for COPD, salt corticosteroids (e.g., fludrocortisone) for orthostatic hypotension, and low-dose glucocorticoid supplements (≤10 mg/day prednisone or equivalent) for adrenal insufficiency.
  6. Exclusion: Severe vaccine allergy history, use of attenuated live vaccines within 28 days before initial treatment, or anticipated need within 6 months after the last dose of the investigational drug.
  7. Uncontrolled systemic diseases, including cardiovascular diseases, organ failure, diabetes, and poorly controlled hypertension.
  8. Unmanageable mental illness or significant medical history that may increase risks or interfere with results.
  9. Thrombotic events within the first 6 months before initial treatment, unless anticoagulation can be discontinued during the screening period.
  10. Irreversible electrolyte imbalances.
  11. Severe infection in the first month before initial treatment, poorly controlled infection, or requiring antibiotic treatment within the past week (excluding prophylactic use).
  12. Pregnant or lactating subjects.
  13. Factors judged by the investigator that may necessitate premature study termination, such as non-compliance, other severe diseases requiring concurrent treatment, severe laboratory abnormalities, or family/social factors affecting subject safety or data/sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AE and SAE | Throughout the whole clinical trial, around 2 years.
  Evaluating the incidence rates of Adverse Events and Serious Adverse Events
DLT | 2 months
  Dose-limiting toxicity.Referencing the results of the exploratory clinical study of ZSNeo-DC1.1 injection, clinical trial outcomes of similar drugs, and the NCI CTCAE 5.0 toxicity assessment criteria to determine DLT. The observation period for DLT is set during the activation of the subject's anti-tumor immune response, from the first day of treatment until 21 days after the third injection.

SECONDARY OUTCOMES:
Assessment of ORR (Objective Response Rate) | For Sequence A/B, ORR is measured both on Day57, and after, ORR is measured when every 8 weeks, until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According toRANO2.0, to assess the proportion of subjects achieving complete remission (CR) or partial remission (PR).
Assessment of DCR (Disease Control Rate) | For Sequence A/B, DCR is measured both on Day57, and after, ORR is measured when every 8 weeks, until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RANO2.0, to assess the proportion of subjects achieving complete remission (CR), partial remission (PR), and stable disease (SD)
Assessment of CBR (Clinical Benefit Rate) | For Sequence A/B, CBR is measured until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RANO2.0, to assess the proportion of subjects in each treatment group with the best overall therapeutic effect, defined as the sum of Complete Remission (CR), Partial Remission (PR), and Stable Disease (SD), lasting for at least 6 months.
Assessment of PFS (Progression Free Survival) | For Sequence A/B, PFS is measured both on Day57, and after, PFS is measured when every 8 weeks), until the date of disease progression or death, whichever came first, assessed up to 2 years.
  According to RANO2.0, to assess the PFS of the patients.
OS (Overall survival) | 2 years
  Time from enrollment to the dates of death from any cause or last follow up reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No